CLINICAL TRIAL: NCT05020977
Title: Physical Actitvity and Blood Pressure Among Ambulance Personnel During Work and Leisure
Status: Completed | Type: Observational
Sponsor: Jonkoping University (Other)
Responsible Party: Principal Investigator, Eleonor Fransson, Associate Professor, Jonkoping University
Other Study IDs: JU 2020/4878-51
Record Dates: First submitted 2021-05-04; First posted 2021-08-25 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Blood Pressure; Work-Related Condition
MeSH Terms: interventions — Blood Pressure; Exercise; Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood pressure, physical activity, health — Observational study of work environment, leisure time, blood pressure, physical activity and health

SUMMARY:
The aim is to describe physical activity and blood pressure during work and leisure time among Swedish ambulance personnel, and to relate this to work- and lifestyle factors.

DETAILED DESCRIPTION:
The work environment for ambulance personnel consists of several factors that might have negative effect on health, for example shift work, long working hours, stress and physical demanding work. Associations between these work-related factors and increased risk of disease, for example cardiovascular- and musculoskeletal disease, have been observed in several studies. However, few studies have specifically been focusing on ambulance personnel.

There is lack of knowledge regarding how work environment factors affect physical activity during work and leisure time among ambulance personnel. Further, the knowledge about blood pressure during work and leisure time is limited for this group.

ELIGIBILITY:
Inclusion Criteria:

* Employed in the ambulance organisation at the time for data collection

Exclusion Criteria:

* Managers and administrative personnel in the ambulance organisation

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses and paramedics employed in the ambulance organisation.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 48 hours
  Ambulatory blood pressure, Objectively measured

SECONDARY OUTCOMES:
Physical activity | 7 days
  Objectively measured with accelerometry
Recovery | baseline, pre-intervention/procedure/surgery
  Self-reported
Health | baseline, pre-intervention/procedure/surgery
  Subjective overall health

CONTACTS AND LOCATIONS:
Overall Officials: Eleonor I Fransson, PhD, Principal Investigator — Jonkoping University
Locations (1):
- Jonkoping University, School of Health and Welfare, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No